CLINICAL TRIAL: NCT02764957
Title: Effects of Green Coffee Extract Supplementation on Anthropometric Measurements, Glycemic Control, Blood Pressure, Lipid Profile
Brief Title: Green Coffee Extract and Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Dr Azita Hekmatdoost, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NationalNFTI
Record Dates: First submitted 2016-05-01; First posted 2016-05-06 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Active Comparator): 400 mg green coffee extract capsules twice per day for 8 weeks The Green coffee extract is standardised with 45% total chlorogenic acid by HPLC
  Interventions: Dietary Supplement: green coffee extract
- control (Placebo Comparator): placebo capsules twice per day for 8 weeks have identical appearance to Green coffee extract capsules and contain starch
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: green coffee extract
  Arms: intervention
Dietary Supplement: placebo
  Arms: control

SUMMARY:
Metabolic syndrome (Mets) is an assemblage of risk factors which can increase the risk of developing type 2 diabetes mellitus and cardiovascular disease. Green coffee extract (GCE) is derived from unroasted coffee beans and has substantial amounts of polyphenols primarily chlorogenic acids (CGA). It has been shown that GCE and CGA can exert a positive influence over Mets components including blood pressure, blood glucose, inflammation, oxidative stress, insulin resistance and blood lipids. Up to our knowledge no study has been conducted on humans in the field of GCA influences on Mets patients. Therefore, this study is planned to evaluate GCA supplementation effects on anthropometric measurements, glycemic control, blood pressure, lipid profile in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference>102 cm in men and >88 cm in women
* Fasting blood glucose>100 mg/dL (5.6 mmol /L)
* Systolic blood pressure>130 mmHg or diastolic blood pressure>85mmHg
* Triglycerides> 150 mg/dL (1.7 mmol/L)

Exclusion Criteria:

* Insulin administration
* Pregnancy and breastfeeding
* regular consumption of coffee and green tea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose | 8 weeks

SECONDARY OUTCOMES:
HOMA-IR | 8 weeks
blood pressure | 8 weeks
insulin | 8 weeks
hemoglubin A1c | 8 weeks
triglyceride | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided